CLINICAL TRIAL: NCT00870246
Title: Influence of Diaphragmatic Mobility on the Exercise Capacity and Dyspnoea in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Diaphragmatic Mobility and Chronic Obstructive Pulmonary Disease
Acronym: DMCOPD
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Celso Ricardo Fernandes de Carvalho, University of Sao Paulo
Other Study IDs: 914/04
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; pulmonary emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: High mobility
- 2: Lower mobility

SUMMARY:
The purpose of this study is to evaluate the influence of diaphragm mobility on exercise capacity and dyspnoea in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is characterized by progressive obstruction of the airways which is partially irreversible. COPD patients commonly present increased resistance to airflow, air trapping, and pulmonary hyperinflation that alters the chest wall placing the respiratory muscles in mechanical disadvantage, thereby increasing both respiratory drive and the sensation of dyspnoea. Furthermore, to prevent dyspnoea, COPD patients reduce their daily living activities leading to loss of physical condition, social isolation, depression and anxiety,whilst compromising their quality of life.

Forced expiratory volume in one second (FEV1) is the main parameter used to establish the severity of pulmonary impairment and disease progression.

Nevertheless, some studies have suggested that FEV1 does not adequately reflect the clinical manifestations of the disease and is only weakly associated with the severity of dyspnoea, health related quality of life (HRQOL) features, and the ability to perform activities of daily living.

Moreover, FEV1 appears not to be a predictor of mortality in COPD patients. Pulmonary hyperinflation has been related with adaptation in diaphragm muscle maintaining the muscle's capacity to generate power whilst reducing its displacement. The importance of the diaphragm in lung mechanics associated with hyperinflation has been the subject of frequent discussion owing to widespread use of lung volume reducing surgery which results in increased movement range of the diaphragm muscle. However, to date, the relationship between diaphragm mobility and functional capacity in COPD patients remains unknown.

The objective of the present study was to evaluate the influence of diaphragm mobility in the exercise capacity and dyspnoea of patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic obstructive pulmonary disease clinically stable (no respiratory crises or hospitalizations within the 30 days preceding the study outset)
* patients receiving optimized clinical medical treatment

Exclusion Criteria:

* patients suffering from other cardiorespiratory diseases
* patients with oxygen-dependent for any reason
* patients classified as obese or as underweight
* patients presenting other respiratory diseases or pleural scars on chest X-rays

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients with moderate or severe COPD were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
spirometer, capacity of exercise, dyspnea | 3 months

SECONDARY OUTCOMES:
diaphragm mobility: the craniocaudal excursion of the intrahepatic branches of the portal vein with the B-mode ultrasound | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Celso Carvalho, professor, Principal Investigator — Sao Paulo University